CLINICAL TRIAL: NCT04496388
Title: The Effect of Different Types of Exercise on Insulin Resistance and Visceral Adipose Tissue in Community Residents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, Principal Investigator, Nurse, ph D student, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 109-035
Record Dates: First submitted 2020-07-25; First posted 2020-08-03 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Exercise, Insulin Resistance, Visceral Adipose Tissue
MeSH Terms: conditions — Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise (Experimental): Aerobic exercise is lasting for nearly 50 minutes each time, including warm-up and stretching for 10 minutes after exercise.
  Interventions: Behavioral: exercise
- Aerobic exercise combined with resistance exercise (Experimental): Aerobic exercise is lasting for nearly 20 minutes each time, and add resistance exercise for 20 minutes. Additional warm-up 10 minutes and stretching for 5 minutes.
  Interventions: Behavioral: exercise
- Aerobic exercise combined with interval training (Experimental): Aerobic exercise is lasting for nearly 20 minutes each time, and add moderal intensity interval training for 10 minutes. Additional warm-up 10 minutes and stretching for 15 minutes.
  Interventions: Behavioral: exercise
- Placebo (Placebo Comparator): No exercise intervention.
  Interventions: Behavioral: No exercise intervention

INTERVENTIONS:
Behavioral: exercise — different type of exercise
  Arms: Aerobic exercise; Aerobic exercise combined with interval training; Aerobic exercise combined with resistance exercise
Behavioral: No exercise intervention — No exercise intervention
  Arms: Placebo

SUMMARY:
Background: Exercise has been proven to effectively reduce incidence of diabetes mellitus and metabolic syndrome. However, there is controversial data from prior studies to inform the type of exercise training recommendations.

Aim: The aim of this study will determine the differences of different type of exercise in the effects of reducing insulin resistance and visceral adipose tissue for community residents.

Methods: The four-arm randomized controlled trial will conducted in adults aged 40 to 70 years old in Tainan. A total of at least 177 patients will randomly assign to the group of aerobic exercise (AE), aerobic exercise combined with resistance exercise (RE), AE combined with medium intensity interval training, and placebo. The participants in exercise group will received 12 weeks, 3 times per week program, including twice a week intervention guided by the intervenors, and once a week exercise guided by the video at home. All the exercise keeps moderate-intensity by monitoring with 64%-75% of the maximum heart rate. Insulin resistance status will be checked by HOMA index at baseline and at exercise intervention after 12 weeks (HOMA index= insulin μU/mL）× glucose（mmol/L）/22.5).

Relevance to clinical practice: The research findings will help the clinical health works to know which type of exercise is the best choice in reducing insulin resistance and visceral adipose tissue in community residents, and can be promoted to the general public to reduce the prevalence of metabolic syndrome as well as prevent the root causes of ill health.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 40 to 70 years old.
* without regular exercise in the past six years.

Exclusion Criteria:

* recent unstable condition involving stroke or those with heart disease, handicap, pregnancy, mental disorders, systolic BP > 200 mmHg, or diastolic BP >110 mmHg.
* those with contraindications in body composition analyzer measurement including people with pacemakers, artificial metal joints, amputated hands or feet, and those who cannot be cooperated with standing during testing.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
visceral adipose tissue | time before intervention(T0) and after 12-weeks exercise intervention (T1)
  measured by the body composition analyzer, which uses bioelectrical impedance analysis to estimate body composition.
insulin resistance | time before intervention(T0) and after 12-weeks exercise intervention (T1)
  Blood samples.Insulin resistance status will be checked by HOMA index at baseline and at exercise intervention after 12 weeks (HOMA index= insulin （μU/mL）× glucose（mmol/L）/22.5). The insulin level and fasting sugar from blood sample will be checked to calculate the insulin resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Hsuan Chang, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang YH, Shun SC, Chen MH, Chang YF. Feasibility of Different Exercise Modalities for Community-Dwelling Residents With Physical Inactivity: A Randomized Controlled Trial. J Nurs Res. 2023 Dec 1;31(6):e301. doi: 10.1097/jnr.0000000000000578. PMID 37883059